CLINICAL TRIAL: NCT00126555
Title: A Phase II Study of ZD1839 and Radiation in Patients With Squamous Cell Carcinoma of the Skin
Brief Title: Gefitinib in Treating Patients Who Are Undergoing Surgery and/or Radiation Therapy for Locally Advanced or Recurrent Squamous Cell Skin Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02893; 2004-0204
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Skin Cancer; Squamous Cell Carcinoma of the Skin
Keywords: squamous cell carcinoma of the skin; recurrent skin cancer; non-melanomatous skin cancer; Radiation; ZD1839; Iressa; Gefitinib
MeSH Terms: conditions — Skin Neoplasms | interventions — Gefitinib; Radiotherapy; Radiation; Surgical Procedures, Operative; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratum I (Gefitinib, Radiotherapy, Surgery) (Experimental): Resectable Strata: Induction Gefitinib (60 days), Surgery followed 3-6 weeks later by daily Radiotherapy 5 days a week for approximately 6-7 weeks then after 4 weeks restart Maintenance Gefitinib for up to additional 12 months post radiation.
  Gefitinib Induction Phase starting dose 250 mg/day, possible doubling to 500 mg/day for no response Day 15; Maintenance dose post radiation starts at same dose level as last dosing of Induction Phase.
  Interventions: Drug: Gefitinib; Radiation: Radiotherapy; Other: laboratory biomarker analysis
- Stratum II (Gefitinib, Radiotherapy/Surgery) (Experimental): Unresectable Strata: Concomitant Radiation/Gefitinib and post-radiation (or post-surgery if surgery is indicated) Gefitinib. Daily Radiotherapy 5 days a week for approximately 6-7 weeks concurrent with Maintenance Gefitinib dose daily up to 12 months.
  Gefitinib Induction Phase starting dose 250 mg/day, possible doubling to 500 mg/day for no response Day 15; Maintenance dose post radiation starts at same dose level as last dosing of Induction Phase.
  Interventions: Drug: Gefitinib; Radiation: Radiotherapy; Procedure: Conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Gefitinib — Oral Gefitinib induction therapy given daily for 2 months at 250 mg/day, once a day for 30 days (1 cycle = 30 days) with at least 2 cycles of treatment (60 days) given. After 2 months evaluate for clinical response (15 days) and resectability (60 days). If after 15 days with no tumor response, daily dose doubled (500 mg), and discontinuation if tumor progression.
  Other Names: Iressa; ZD 1839
Radiation: Radiotherapy — Undergo radiation therapy treatments once a day Monday through Friday for about 7 weeks. Each treatment takes about 15 minutes.
  Other Names: irradiation; therapy, radiation
Procedure: Conventional surgery — Undergo surgery
  Other Names: surgery, conventional
  Arms: Stratum II (Gefitinib, Radiotherapy/Surgery)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The goal of this clinical research study is to learn if giving Iressa (Gefitinib or ZD1839) with surgery and/or radiation will help to control squamous cell carcinoma of the skin. The safety of this treatment will also be studied

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Early progression rate (progression during ZD1839 induction).

II. Feasibility of induction ZD1839 (for all patients) and concomitant ZD1839 with radiotherapy (for unresectable patients).

III. Toxicities of induction ZD1839 (for all patients) and concomitant ZD1839 with radiotherapy (for unresectable patients).

SECONDARY OBJECTIVES:

I. Response: clinical responses to induction therapy.

II. Failures: frequency and timing of local and distant failures.

III. Biomarkers: biomarker levels in tumor and normal tissue.

TERTIARY OBJECTIVES:

I. For progressive disease responders, patients will be followed for locoregional and distant metastases data.

II. Feasibility of maintenance ZD1839.

III. Toxicities of maintenance ZD1839.

OUTLINE: Patients are assigned to 1 of 2 groups.

STRATUM I (initially resectable tumor): Patients undergo radiotherapy once daily (QD) 5 days a week for approximately 6-7 weeks. Patients also receive gefitinib orally (PO) QD for up to 12 months

STRATUM II (initially unresectable tumor): Patients undergo radiotherapy QD 5 days a week for approximately 6-7 weeks. Patients also receive concurrent gefitinib PO QD for 6-7 weeks. Patients then undergo surgery. After surgery, patients receive gefitinib PO QD for up to 12 months.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Within 12 weeks (+/- 2 weeks) prior to study entry, patients must have histologically or cytologically confirmed squamous cell carcinoma (SCC) of skin that is either locally advanced or recurrent with measurable disease; if the biopsy was collected outside of MDACC, the MDACC Pathology Department must assess and confirm the SCC diagnosis
* Patients may have previous surgical intervention with residual or recurrent disease
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm*3
* Total bilirubin within normal institutional limits
* aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) =< 2.5 * institutional upper limit of normal
* Creatinine within normal institutional limits OR; creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Tumors must be at least 2 cms in size or have histological or cytological verification of muscle, bone, lymph node metastasis, or perineural involvement, as measured by the treating physician(s) or National principal investigator (PI)
* Negative serum pregnancy test for women of child-bearing potential (performed within 14 days, +/- 1 day, prior to start of treatment); women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in the study, she should inform her treating physician(s) immediately
* Ability to understand and the willingness to sign a written Informed Consent Document (ICD); in the event that non-English speaking participants are eligible for this study, a short form (if applicable) or an ICD in their language, will be utilized and completed in accordance with the MD Anderson's "Policy For Consenting Non-English Speaking Participants"

Exclusion Criteria:

* Patients who have previous radiotherapy to the proposed site of skin cancer
* Patients with active cancers other than skin
* Patients currently receiving any other investigational agents at time of study enrollment; patients may have received investigational agents in the past; no washout time period is required
* Patients with a history of brain metastases must be excluded from this clinical study because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZD1839
* Age less than 18 years
* Presence of uncontrolled intercurrent illness (co-morbid conditions) that would limit compliance with study requirements including , but not limited to, ongoing or active infection requiring parenteral antibiotics at time of study registration, symptomatic congestive heart failure (NYHA class II or greater), unstable angina pectoris or cardiac arrhythmia requiring maintenance medication
* Pregnant women are excluded from this study because ZD1839 is a signal transduction inhibitor agent with the potential for teratogenic or abortifacient effects; there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ZD1839, breastfeeding should be discontinued if the mother is treated with ZD1839
* Patients with known immune deficiency are at an increased risk when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded due to the possible pharmacokinetic interactions with ZD1839; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* CYP3A4 inducing agents; patients receiving the following CYP3A4 inducing agents will be excluded; these include: carbamazepine, ethosuximide, griseofulvin, modafinil, nafcillin, oxcarbazepine, Phenobarbital, phenylbutazone, phenytoin, rifampin, rifabutin, St. John's Wort, and sulfinpyrazone
* Patients with distant metastatic disease as determined by diagnostic imaging (i.e., chest x-rays) and/or hematologic assessments (i.e., liver enzymes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randal Weber, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Web Site — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 08, 2005 to March 13, 2008. All participants were recruited at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 23 participants enrolled, one participant who was not evaluable for response withdrew before beginning treatment and is included the study demographics.
Groups:
- Gefitinib, Radiotherapy, Surgery: Gefitinib Induction therapy daily for 2 months then evaluated for clinical response and resectability: Resectable strata who have achieved at least stable disease receive surgery followed by radiation treatment, if indicated, and 12 additional months of Gefitinib post radiation. Unresectable strata who have achieved at least stable disease receive concomitant radiation/Gefitinib and 12 additional months of Gefitinib post-radiation (or post-surgery if surgery is indicated). Maintenance Phase of Gefitinib starts at same dose level as last dosing of Induction phase.
Period: Overall Study
Arm/Group | Gefitinib, Radiotherapy, Surgery
Started | 23
Stratum 1- Resectable | 18 (1 participant did not participate)
Stratum 2- Unresectable | 4
Completed | 17
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Not completed — Progressive Disease | 3

BASELINE CHARACTERISTICS:
Population: Of the 23 participants enrolled, one participant who was not evaulable for response withdrew before beginning treatment.
Arm/Group | Gefitinib, Radiotherapy, Surgery
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] — Demographics are reported as consolidated information for both stratum.
  years | 65 [27 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Early Progression Rate
Description: Number of participants out of total participants with progression following two 30 day courses of Gefitinib. Tumor response evaluated by Response Evaluation Criteria in Solid Tumors by physical exam, computed tomography (CT) or Magnetic Resonance Imaging (MRI). Progressive disease defined as determined as response to Gefitinib induction therapy: Progression: 25% increase in sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer). Participants restaged on days 15 and 60 of treatment.
Time Frame: Baseline to 60 days, up to 2 courses of induction therapy
Measure: Number; unit: percentage of participants
Groups:
- Gefitinib, Radiotherapy, Surgery: Gefitinib Induction therapy daily for 2 months then evaluated for clinical response and resectability: Resectable strata who have achieved at least stable disease receive surgery followed by radiation treatment, if indicated, and 12 additional months of Gefitinib post radiation. Unresectable strata who have achieved at least stable disease receive concomitant radiation/Gefitinib and 12 additional months of Gefitinib post-radiation (or post-surgery if surgery is indicated). Maintenance Phase of Gefitinib starts at same dose level as last dosing of Induction phase.
  Gefitinib Induction Phase starting dose 250 mg/day, possible doubling to 500 mg/day for no response Day 15; Maintenance dose post radiation starts at same dose level as last dosing of Induction Phase.
Arm/Group | Gefitinib, Radiotherapy, Surgery
Number analyzed (Participants) | 22
percentage of participants | 31.8

2. Primary Outcome: Number of Participants With Response Rate During Induction, Dose Escalation, and Concomitant With Radiation.
Description: Completion Induction phase, participants are evaluated for clinical response and resectability. Resectable participants who had achieved at least stable disease and received surgery followed by radiation. Unresectable participants who had achieved at least stable disease received concomitant radiation/Gefitinib.
Time Frame: Up to 100 days
Measure: Count of Participants; unit: Participants
Groups:
- Patients Completed Induction Gefitinib: All patients treated induction gefitinib within 60 days
- Patients Received the Escalated Gefitinib Dose: Patients treated induction gefitinib evaluated as Stable Disease at 15 days, patients received the escalated gefitinib dose for 45 days, total of 60 days.
- Patients Treated Radiation and Concurrent Gefitinib: Unresectable patients treated concomitant gefitinib with radiotherapy
Arm/Group | Patients Completed Induction Gefitinib | Patients Received the Escalated Gefitinib Dose | Patients Treated Radiation and Concurrent Gefitinib
Number analyzed (Participants) | 17 | 6 | 3
Participants
  Complete Response (CR) | 4 | 1 | 0
  Partial Response (PR) | 5 | 0 | 2
  Stable Disease (SD) | 5 | 3 | 1
  Progressive Disease (PD) | 3 | 2 | 0

3. Primary Outcome: Toxicity as Assessed by the National Cancer Institute (NCI) Common Toxicity Criteria Associated With Gefitinib Therapy: Expected Toxicities (Grade 1 - 3)
Description: Severity and timing of toxicities evaluated according to NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 3. Occurrences of late (post-radiation) toxicities that are radiation-related monitored and included.
Time Frame: Up to 5 years
Population: Of 23 enrolled, 1 withdrew, 2 went off study during induction for adverse events and 3 had progressive disease. Of 17 continuing to clinical response assessment (11 on 250 mg/day Induction dose & 6 to 500 mg/day dose escalation), 12 were resectable (2 refused), 2 unresectable and 3 had disease progression leaving only 6 for maintenance.
Measure: Number; unit: participants
Groups:
- Induction Phase: Participants received Gefitinib Induction therapy daily for 2 months then were evaluated for clinical response and resectability: Gefitinib Induction Phase dose 250 mg/day with no doubling for no response at Day 15.
- Induction With Dose Escalation: Participants received Gefitinib Induction therapy daily for 2 months then were evaluated for clinical response and resectability: Gefitinib starting dose 250 mg/day with doubling to 500 mg/day for no response Day 15.
- Radiation With Gefitinib: Participants received Radiation with Gefitinib therapy following evaluation for clinical response and resectability at Induction (with or without dose doubling): Resectable strata who achieved at least stable disease received surgery followed by radiation treatment and 12 additional months of Gefitinib post radiation; and the Unresectable strata who achieved at least stable disease received concomitant radiation/Gefitinib and 12 additional months of Gefitinib post-radiation (or post-surgery if surgery is indicated).
- Maintenance: Maintenance Phase of Gefitinib starts at same dose level as last dosing of Induction phase (Gefitinib Induction dose 250 mg/day or 500 mg/day dose escalation).
Arm/Group | Induction Phase | Induction With Dose Escalation | Radiation With Gefitinib | Maintenance
Number analyzed (Participants) | 11 | 6 | 17 | 6
participants
  Fatigue | 11 | 5 | 3 | 2
  Dry skin | 2 | 2 | 1 | 3
  Pruitis | 4 | 2 | 0 | 1
  Rash/desquamation | 4 | 2 | 1 | 1
  Rash/acneiform | 7 | 4 | 2 | 4
  Anorexia | 1 | 2 | 3 | 3
  Diarrhea | 10 | 0 | 0 | 6
  Nausea | 6 | 1 | 3 | 0
  Vomiting | 3 | 0 | 1 | 0
  Elevation of alanine transferase (ALT) | 3 | 2 | 0 | 0
  Elevation of asparagine transferase (AST) | 4 | 2 | 1 | 1
  Elevation of Creatinine | 2 | 0 | 0 | 0
  Abdominal pain | 2 | 0 | 0 | 1
  Dry eyes | 1 | 0 | 1 | 0
  Ocular/visual, other | 0 | 1 | 0 | 0

4. Primary Outcome: Toxicity as Assessed by the National Cancer Institute (NCI) Common Toxicity Criteria Associated With Gefitinib Therapy: UnExpected Toxicities (Grade 1 - 3)
Description: as for outcome 3
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Induction Phase With Dose Escalation: Participants received Gefitinib Induction therapy daily for 2 months then were evaluated for clinical response and resectability: Gefitinib starting dose 250 mg/day with doubling to 500 mg/day for no response Day 15.
- Maintenance Phase: Maintenance Phase of Gefitinib starts at same dose level as last dosing of Induction phase (Gefitinib Induction dose 250 mg/day or 500 mg/day dose escalation).
Arm/Group | Induction Phase | Induction Phase With Dose Escalation | Radiation With Gefitinib | Maintenance Phase
Number analyzed (Participants) | 11 | 6 | 17 | 6
participants
  Allergic reaction | 1 | 0 | 0 | 1
  Anemia | 3 | 1 | 2 | 3
  Weight Loss | 1 | 0 | 1 | 1
  Alopecia | 0 | 0 | 1 | 1
  Taste alteration | 1 | 0 | 0 | 0
  Epistaxis | 1 | 0 | 0 | 0
  Infection | 0 | 1 | 0 | 0
  Elevated BUN | 1 | 0 | 0 | 1
  Elevated White Blood Cell Count (CBC) | 1 | 0 | 0 | 0
  Blurred vision | 1 | 0 | 1 | 1
  Insomnia | 0 | 0 | 0 | 1
  Depression | 0 | 0 | 0 | 1
  Tooth pain | 1 | 0 | 0 | 0

5. Secondary Outcome: Clinical Response According to Response Evaluation Criteria In Solid Tumors (RECIST)
Description: Number participants with response defined by RECIST: Complete Response (CR): Disappearance all disease; No new lesions/non-evaluable disease; Responders on none/only maintenance doses of corticosteroids. Partial Response (PR): >/= 50% decrease under baseline in sum products perpendicular diameters of measurable lesions; No progression evaluable disease/new lesions; Responders on same/decreasing doses dexamethasone & stable/improved neurological exams. Stable/No Response (SD): Not qualify for CR, PR, or progression; requires minimum 12 weeks duration; Responders on same/decreasing doses dexamethasone & stable/improved neurological exams. Progression (PD): 25% increase in sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease), OR clear worsening any evaluable disease, OR appearance any new lesion/site, OR failure to return due to death/deteriorating condition. All measurable/evaluable sites assessed using same baseline techniques.
Time Frame: Up to 5 years
Population: One participant of 23 enrolled withdrew prior to treatment.
Measure: Number; unit: participants
Arm/Group | Gefitinib, Radiotherapy, Surgery
Number analyzed (Participants) | 22
participants
  Complete Response (CR) | 4
  Partial Response (PR) | 6
  Stable Disease (SD) | 5
  Progressive Disease (PD) | 7

6. Secondary Outcome: Frequency and Timing of Local and Distant Failures
Time Frame: From study entry to first documented local recurrence or last patient contact, assessed up to 5 years
Population: Two participants did not complete study treatment (Surgery + Radiotherapy) of 17 progressed and was removed from the study.
Measure: Number; unit: participants
Groups:
- Recurrence Status: Patients had recurrence within the first year after completion of treatment
- Survival Status: At the time of last contact
Arm/Group | Recurrence Status | Survival Status
Number analyzed (Participants) | 15 | 15
participants
  Local recurrence | 2 | 0
  unknown | 1 | 5
  Dermal metastases | 0 | 0
  No Evidence of Disease (NED) | 12 | 5
  Living with disease | 0 | 0
  Died of their disease (DOD) | 0 | 2
  Died from other causes | 0 | 3

7. Other Pre Specified Outcome: Change in Epidermal Growth Factor Receptor (EGFR) and Phospho-Akt Expression
Description: Samples were not available from all participants because the protocol specified that consenting to tissue biopsies was optional. In addition, some participants presented with regional recurrences, which were not superficially accessible. The sample size was too small to determine the EGFR-proliferative responses activated by the AKT pathway; hence, the monitoring of the status of activated phospho-AKT as an independent marker of EGFR activation could not be performed.
Time Frame: Baseline
Population: Samples were not available from all participants because the protocol specified that consenting to tissue biopsies was optional. Sample size was too small to determine EGFR-proliferative responses activated by the AKT pathway;hence, monitoring of the status of activated phospho-AKT as an independent marker of EGFR activation could not be performed.
Arm/Group | Gefitinib, Radiotherapy, Surgery
Number analyzed (Participants) | 0

8. Post Hoc Outcome: Participant Treatment Following Induction Therapy
Description: Treatment received following two 30-day cycles (60 days) of 250 mg gefitinib given by mouth daily. Participant treatment reported as percentage of total treated participants out of total treated.
Time Frame: Following 60 days of Gefitinib induction treatment
Measure: Number; unit: percentage of participants
Arm/Group | Gefitinib, Radiotherapy, Surgery
Number analyzed (Participants) | 22
percentage of participants
  Surgery Alone | 11.8
  Definitive Radiation | 17.6
  Radiation and Concurrent Gefitinib | 11.8
  Surgery, Post-Op Radiation & Concurrent Gefitinib | 47

ADVERSE EVENTS:
Time Frame: Adverse event reporting up to 30 days after last dose investigational agent, up to 12 months following radiotherapy. Active study period June 2005 to September 2008.
Description: One participant in Stratum I out of total 23 enrolled participants withdrew prior to any treatment and is not included in adverse event reporting.
Groups:
- Gefitinib, Radiotherapy, Surgery: Resectable Strata: Induction Gefitinib (60 days), Surgery followed 3-6 weeks later by daily Radiotherapy 5 days a week for approximately 6-7 weeks then after 4 weeks restart Maintenance Gefitinib for up to additional 12 months post radiation.
  Unresectable Strata: Concomitant Radiation/Gefitinib and post-radiation (or post-surgery if surgery is indicated) Gefitinib. Daily Radiotherapy 5 days a week for approximately 6-7 weeks concurrent with Maintenance Gefitinib dose daily up to 12 months.
  Gefitinib Induction Phase starting dose 250 mg/day, possible doubling to 500 mg/day for no response Day 15; Maintenance dose post radiation starts at same dose level as last dosing of Induction Phase.
Arm/Group | Gefitinib, Radiotherapy, Surgery
Serious Adverse Events (participants affected / at risk) | 5/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib, Radiotherapy, Surgery (N=22)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 2 — Grade 3
Confusion (Nervous system disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Depression (Nervous system disorders) | 1
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 5
Diarrhea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Cardiac disorders) | 1
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 2
Insomnia (General disorders) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Pain of skin, Ear (Ear and labyrinth disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Tumor Pain (General disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib, Radiotherapy, Surgery (N=22)
Abdominal pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 5
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 3
Allergic reaction (Immune system disorders) | 2
Allergic rhinitis (Immune system disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 13
Anorexia (Gastrointestinal disorders) | 6
Anxiety (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 10
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
White Blood Count Elevated (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Metabolism and nutrition disorders) | 2
Blurred vision (Eye disorders) | 3
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 1
Conjunctivitis (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Metabolism and nutrition disorders) | 4
Dehydration (Gastrointestinal disorders) | 1
Depression (Nervous system disorders) | 2
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 3
Diarrhea (Gastrointestinal disorders) | 15
Dizziness (Nervous system disorders) | 3
Dry eye (Eye disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 6
Dysgeusia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Ear Pain/Pressure (Ear and labyrinth disorders) | 2
Edema face (Skin and subcutaneous tissue disorders) | 4 — Face (2), Limbs (2)
Epistaxis (General disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
External ear pain (Ear and labyrinth disorders) | 2
Eye Erythema Irritation (Eye disorders) | 3 — Keratitis and Erythema
Eye Pain (Eye disorders) | 1
Facial pain (General disorders) | 3
Fatigue (General disorders) | 13
Fever (General disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
General disorders and administration site conditions (General disorders) | 3 — FALL, PRESYNCOPAL SYMPTOMS, GENERALIZED BODY ACHES
Gingival pain (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Cardiac disorders) | 7
Hyperuricemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypothyroidism (Metabolism and nutrition disorders) | 1
Infection (Infections and infestations) | 2
Insomnia (General disorders) | 1
BUN Elevation/Change (Investigations) | 7
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nail loss (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 13
Oral Pain (Gastrointestinal disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Photophobia (Eye disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash acneiform (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Rectal pain (Gastrointestinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Tumor pain (General disorders) | 7
Urinary tract infection (Renal and urinary disorders) | 1
Urticaria (Immune system disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (General disorders) | 4
White blood cell decreased (Blood and lymphatic system disorders) | 1
Wound dehiscence (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less